CLINICAL TRIAL: NCT05389319
Title: A Phase Ia, Dose-finding Study to Assess the Safety and Immunogenicity of an Orf Virus-based COVID-19 Vaccine Booster (Prime-2-CoV_Beta) in Healthy Adults
Brief Title: A Study to Assess the Safety and Immunogenicity of a COVID-19 Vaccine Booster in Healthy Adults
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The clinical trial was temporarily suspended to account for investigating IMP quality aspects.
Sponsor: University Hospital Tuebingen (Other)
Collaborators: FGK Clinical Research GmbH (Industry); VisMederi srl (Industry); Staburo GmbH (Industry); Viedoc Technologies AB (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PRiME2_21_1
Record Dates: First submitted 2022-05-24; First posted 2022-05-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: COVID-19; vaccine; Orf virus; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — PRIME-2-CoV_Beta COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Cohorts 1 to 5 will include a safety lead with 1 sentinel participant. If no safety issues occurred within the on-site monitoring period as assessed by the investigator and solicited during telephone visits, the next 2 participants in that dose cohort will be vaccinated. After an 48-hour observation period and assuming no safety issues were identified in these 2 participants, an additional 4 participants will be vaccinated. After a 48-hour observation period, and assuming that no safety problems were noted in these 4 participants, the remaining participants in the dosing group will be vaccinated. Each participant will be observed for at least 4 hours at the study center after Prime-2-CoV_Beta booster vaccination. After the last participant of each of the Cohorts 1 to 4 has completed 7 days of follow up after the Prime-2-CoV_Beta booster vaccination, all safety data will be reviewed by the safety review committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1 (Experimental): Prime-2-CoV_Beta, dose: 30 000 PFUs
  Interventions: Biological: Prime-2-CoV_Beta
- Cohort 2 (Experimental): Prime-2-CoV_Beta, dose: 300 000 PFUs
  Interventions: Biological: Prime-2-CoV_Beta
- Cohort 3 (Experimental): Prime-2-CoV_Beta, dose: 3 000 000 PFUs
  Interventions: Biological: Prime-2-CoV_Beta
- Cohort 4 (Experimental): Prime-2-CoV_Beta, dose: 150 000 000 PFUs
  Interventions: Biological: Prime-2-CoV_Beta
- Cohort 5 (Experimental): Prime-2-CoV_Beta, dose: 30 000 000 PFUs
  Interventions: Biological: Prime-2-CoV_Beta

INTERVENTIONS:
Biological: Prime-2-CoV_Beta — 1 intramuscular injection (1.0 mL each) into the deltoid muscle on Day 1

SUMMARY:
This is an open-label, first-in-human, dose-finding study to evaluate the safety and immunogenicity of a booster vaccination of Prime-2-CoV_Beta in healthy participants who had received the full course of vaccination, including booster vaccination (i.e., having received 3 doses) with the Pfizer/BioNTech-BNT162b2 vaccine (Comirnaty).

DETAILED DESCRIPTION:
Eligible participants will undergo baseline assessments and will receive 1 injection of Prime-2-CoV_Beta at Day 1. Participants will be followed up through 6 months post-booster vaccination. Follow-up visits will be performed at Days 4, 8, 15, 29, and Months 3 and 6, to assess the safety, tolerability, and immunogenicity of Prime-2-CoV_Beta. Additional safety and tolerability data will be assessed 1 day and 2 days after booster vaccination (Days 2 and 3) by telephone. A total of 60 participants is planned to be vaccinated in 5 cohorts of 12 participants each. Dose ranging of Prime-2-CoV_Beta will be done by dose escalation with doses ranging from 3x10000 plaque forming units (PFUs) up to 3x10 000 000 PFUs

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria

1. Healthy adult men or women aged 18 to 55 years
2. Full course of vaccination, including booster vaccination (i.e., having received 3 doses) with Comirnaty, with the booster dose being administered at least 10 weeks before Day 1 as documented in a respective vaccination certificate
3. Able to understand the participant information and providing written informed consent
4. Body mass index of 18.5 to 30.0 kg/m² and weight > 50 kg at Screening
5. Women of childbearing potential must:

   1. have a negative pregnancy test at Screening (blood) and at Day 1 (urine)
   2. agree to use, and be able to comply with, highly effective measures of contraception without interruption, from 14 days before Prime-2-CoV_Beta booster vaccination until the end of the study.

   A highly effective method of contraception or birth control (failure rate less than 1% per year when used consistently and correctly) for this study: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal, injectable), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, sexual abstinence or vasectomized sexual partner. Abstinence is only acceptable as true abstinence when this is in line with the preferred and usual lifestyle of the participant (abstinent on a long-term and persistent basis). The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods and withdrawal] are not acceptable methods of contraception.) Postmenopausal (no menses for at least 1 year without alternative medical cause) or surgically sterile women (tubal ligation, hysterectomy or bilateral oophorectomy) may be enrolled.
6. Male participants must agree not to intend to father a child or to donate sperm starting at Screening, throughout the clinical study. Male participants must also

   1. abstain from sexual intercourse with a female partner (acceptable only if it is the participant's usual form of birth control/lifestyle choice: abstinent on a long-term and persistent basis). The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the participant or
   2. use adequate barrier contraception (male condom) during treatment with the investigational product until the end of the study, and
   3. ensure that, if they have a female partner of childbearing potential, the partner uses a highly effective contraceptive method as outlined in inclusion criterion number 5
   4. use condoms during the entire study if they have a pregnant partner, to avoid exposure of the fetus to the investigational product
7. Willing and able to comply with all study procedures based on the investigator's judgment

Exclusion Criteria:

Previous and concomitant therapy:

1. Receipt of any vaccine (licensed or investigational) from 4 weeks before Prime-2-CoV_Beta booster vaccination or anticipated vaccination during the study until 6 weeks after the Prime-2-CoV_Beta booster vaccination
2. Previous vaccination against COVID-19 with vaccines (licensed or investigational) other than Comirnaty
3. Current or previous treatment with another investigational drug and/or medical device (within 30 days of enrollment or 5 half-lives of that investigational drug)
4. Administration of immunoglobulins or any blood products within 2 months of Prime-2-CoV_Beta booster vaccination
5. Chronic administration of medication associated with impaired immune responsiveness as judged by the investigator (including, but not limited to: immunosuppressive therapy, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy shots for hypo-sensitization, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs) within 2 months before the Prime-2-CoV_Beta booster vaccination (Day 1). Inhaled/nebulized, intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.

   Previous and concomitant medical condition:
6. Active SARS-CoV-2 infection, confirmed by a commercially available SARS-CoV-2 rapid antigen test at Day 1, or currently on quarantine
7. Confirmed (by real-time quantitative polymerase chain reaction) SARS-CoV-2 infection after 2nd vaccination with Comirnaty
8. Known history of severe adverse reactions to any vaccine and/or severe allergic reactions to any component of the study vaccine, to any drug, or to any other exposure
9. Known history of angioedema
10. Pregnant or lactating women
11. Any confirmed or suspected immunosuppressive or immunodeficient condition
12. Known history of Guillain-Barré Syndrome
13. Known infection with human immunodeficiency virus, hepatitis C virus or hepatitis B virus
14. Active cancer (malignancy) within 5 years before Day 1 (except for adequately treated non-melanomatous skin carcinoma, at the discretion of the investigator)
15. Moderate or severe illness and/or fever > 38.0 °C within 1 week before Prime-2-CoV_Beta booster vaccination
16. Any clinically significant health problem (medical history and physical examination) or clinically significantly abnormal finding in biochemistry and/or hematology blood tests, urinalysis, or electrocardiogram at Screening according to the investigator's opinion
17. Current or history of cardiovascular disease or structural cardiac disease (including chronic or congenital heart conditions, such as chronic hypertension, coronary heart disease, myocardial infarction and arrhythmias, hypertrophic cardiomyopathy, as well as a history of myocarditis after mRNA vaccinations)
18. History of mRNA vaccination-associated adverse events that were in nature and severity beyond the common AEs expected
19. Current or history of gastrointestinal disease, liver disease, renal disease or endocrine disorders, (including diabetes) and neurological illness (excluding migraine), when judged as clinically significant according to the investigator's opinion
20. Current or history of chronic respiratory diseases, including mild asthma treated by on-demand medication (resolved childhood asthma is allowed)
21. Current or history of alcohol and/or drug abuse within the last 6 months before Day 1

    Previous and concomitant clinical study experience
22. Current participation in another study or previous enrollment in this clinical study

    Other exclusion criteria
23. Investigator or employee of the study group or sponsor with direct involvement in the proposed study or relatives of the research staff with direct involvement in the proposed study
24. Prolonged exposure to sheep or goats (e.g., shepherds, sheep farmer)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) throughout the study | Day 1 (vaccination day) to month 6 (end of study visit, ±14 days)
  All safety data will be summarized descriptively overall and by cohort. TEAEs will be summarized by descriptive statistics using contingency tables (counts of events, number and proportion of participants with events) and presented by system organ class and preferred term, as well as by severity.
Proportion of participants with solicited local adverse events (first 7 days after Prime-2-CoV_Beta booster vaccination): pain at injection site, redness, induration, and swelling. | Day 1 (vaccination day) to day 8 (Visit 3; ±1 day)
  Solicited local adverse events will be summarized by descriptive statistics using contingency tables (counts of events, number and proportion of participants with events).
Proportion of participants with solicited systemic adverse events (first 7 days after Prime-2-CoV_Beta booster vaccination): fever, fatigue, headache, chills, vomiting, nausea, diarrhea, new or worsened muscle pain, new or worsened joint pain. | Day 1 (vaccination day) to day 8 (Visit 3; ±1 day)
  Solicited systemic adverse events will be summarized by descriptive statistics using contingency tables (counts of events, number and proportion of participants with events).
Proportion of participants with unsolicited treatment-emergent adverse events throughout the study | Day 1 (vaccination day) to month 6 (end of study visit, ±14 days)
  All unsolicited adverse events which occur after the first administration of investigational product are defined as treatment-emergent adverse events. Treatment-emergent adverse events will be summarized by descriptive statistics using contingency tables (counts of events, number and proportion of participants with events) and presented by system organ class and preferred term, as well as by severity.

SECONDARY OUTCOMES:
Level of neutralizing antibody titers versus SARS CoV-2 (Wuhan wild type) at each post-booster vaccination assessment | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Immunogenicity endpoints will be descriptively analyzed by cohort and visit. Separate analyses will be done for the different parameters, e.g., different antibodies evaluated with different serological immunogenicity assays.
Geometric mean fold rise (GMFR) of neutralizing antibodies (versus Wuhan wild type) from Baseline to each post-booster vaccination assessment | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  The fold change from Baseline will be computed for each participant. The fold rise is calculated as the ratio of the post- vs pre-vaccination titer value. The fold change from Baseline will be summarized using descriptive statistics by cohort and visit. Additionally, the GMFR with 95% CI will be presented.
IgG antibody titer versus SARS-CoV-2 receptor-binding protein | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Immunogenicity endpoints will be descriptively analyzed by cohort and visit. Separate analyses will be done for the different parameters, e.g., different antibodies evaluated with different serological immunogenicity assays.
Geometric mean titers (GMT) of receptor-binding protein-specific IgG antibodies | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Immunogenicity endpoints will be descriptively analyzed by cohort and visit. Separate analyses will be done for the different parameters, e.g., different antibodies evaluated with different serological immunogenicity assays.
Geometric mean fold rise of receptor-binding protein-specific IgG antibodies from Baseline | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  The fold change from Baseline will be computed for each participant. The fold rise is calculated as the ratio of the post- vs pre-vaccination titer value. The fold change from Baseline will be summarized using descriptive statistics by cohort and visit. Additionally, the geometric mean fold rise with 95% confidence interval will be presented.
Proportion of participants with adverse events of special interest throughout the study | Day 1 (vaccination day) to day 8 (Visit 3; ±1 day)
  Adverse events of special interest will be summarized by descriptive statistics using contingency tables (counts of events,number and proportion of participants with events) and presented by system organ class and preferred term, as well as by severity.
  The frequency (% of participants) of adverse events of special interest throughout the study will be tabulated.

OTHER OUTCOMES:
IgG antibody titer versus SARS-CoV-2 S1 protein | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Immunogenicity endpoints will be descriptively analyzed by cohort and visit. Separate analyses will be done for the different parameters, e.g., different antibodies evaluated with different serological immunogenicity assays.
Geometric mean titers of IgG S1-specific antibodies | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Absolute values of serological immunogenicity assays as described will be presented using descriptive summary statistics by cohort and visit. Additionally, Geometric mean titers with 95% confidence interval (CI) will be provided. For each cohort, serological immunogenicity assays will be presented graphically displaying Geometric mean titers with 95% CIs at all visits.
Geometric mean fold rise of IgG S1-specific antibodies from Baseline | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  The fold change from Baseline will be computed for each participant. The fold rise is calculated as the ratio of the post- vs pre-vaccination titer value. The fold change from Baseline will be summarized using descriptive statistics by cohort and visit. Additionally, the geometric mean fold rise with 95% CI will be presented.
IgG antibody titer versus SARS-CoV-2 N-protein | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Immunogenicity endpoints will be descriptively analyzed by cohort and visit. Separate analyses will be done for the different parameters, e.g., different antibodies evaluated with different serological immunogenicity assays.
Geometric mean titers of N-specific IgG antibodies | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Absolute values of serological immunogenicity assays as described will be presented using descriptive summary statistics by cohort and visit. Additionally, geometric mean titers with 95% confidence interval (CI) will be provided. For each cohort, serological immunogenicity assays will be presented graphically displaying geometric mean titers with 95% CIs at all visits.
Geometric mean fold rise of N-specific IgG antibodies from Baseline | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  The fold change from Baseline will be computed for each participant. The fold rise is calculated as the ratio of the post- vs pre-vaccination titer value. The fold change from Baseline will be summarized using descriptive statistics by cohort and visit. Additionally, the geometric mean fold rise with 95% confidence intervals will be presented.
Level of neutralizing antibody titers versus the variant of concern SARS-CoV-2_Beta, SARS-CoV-2_Delta and SARS-CoV-2_Omicron at each post-booster vaccination assessment | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  Immunogenicity endpoints will be descriptively analyzed by cohort and visit. Separate analyses will be done for the different parameters, e.g., different antibodies evaluated with different serological immunogenicity assays.
Geometric mean fold rise of neutralizing antibodies from Baseline to each post-booster vaccination assessment | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 3 (±14 days), month 6 (end of study visit, ±14 days)
  The fold change from Baseline will be computed for each participant. The fold rise is calculated as the ratio of the post- vs pre-vaccination titer value. The fold change from Baseline will be summarized using descriptive statistics by cohort and visit. Additionally, the geometric mean fold rise with 95% confidence intervals will be presented.
Percentage of cytokine producing S and N protein-specific T-cells compared to Baseline | Day 1 (vaccination day), day 8 (±1 day), day 15 (±2 days), day 29 (±1 day), month 6 (end of study visit, ±14 days)
  Analyses based on S- and N-specific antibodies will be performed as described for receptor-binding protein specific antibodies.
Additional assays to measure the immune response to Prime-2-CoV_Beta and immune response to the Orf virus vector backbone | Day 1 (vaccination day), day 15 (±2 days), day 29 (±1 day), month 6 (end of study visit, ±14 days)
  Orf virus-specific antibodies will be summarized descriptively as described for virus-specific antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Esen, Dr., Principal Investigator — University Hospital Tübingen, Institute of Tropical Medicine
Locations (2):
- Germany (2):
  - University Hospital Tübingen, Institute of Tropical Medicine, Tübingen, Baden-Wurttemberg
  - Bernhard-Nocht-Institut für Tropenmedizin, Hamburg, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Esen M, Fischer-Herr J, Gabor JJ, Gaile JM, Fleischmann WA, Smeenk GW, de Moraes RA, Belard S, Calle CL, Woldearegai TG, Egger-Adam D, Haug V, Metz C, Reguzova A, Loffler MW, Balode B, Matthies LC, Ramharter M, Amann R, Kremsner PG. First-in-Human Phase I Trial to Assess the Safety and Immunogenicity of an Orf Virus-Based COVID-19 Vaccine Booster. Vaccines (Basel). 2024 Nov 18;12(11):1288. doi: 10.3390/vaccines12111288. PMID 39591190